CLINICAL TRIAL: NCT02754752
Title: Randomized-Controlled Trial of Acupuncture for Chronic Pain After Breast Cancer Treatment
Brief Title: Electroacupuncture Therapy in Reducing Chronic Pain in Patients After Breast Cancer Treatment
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Gateway for Cancer Research (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2015-0750; NCI-2016-00792 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0750 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-04-26; First posted 2016-04-28 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Stage I Breast Cancer AJCC v7; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage III Breast Cancer AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7
MeSH Terms: conditions — Breast Neoplasms | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group I (electroacupuncture therapy) (Experimental): Patients undergo electroacupuncture therapy over 45 minutes 2-3 times per week over 4 weeks for a total of 10 sessions.
  Interventions: Procedure: Electroacupuncture Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (sham electroacupuncture therapy) (Placebo Comparator): Patients undergo modified electroacupuncture therapy over 45 minutes 2-3 times per week over 4 weeks for a total of 10 sessions. Acupuncture needles are placed in different locations using a different technique than those used for Group I.
  Interventions: Procedure: Electroacupuncture Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group III (waitlist control) (Active Comparator): Patients receive standard of care without any kind of acupuncture therapy.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Electroacupuncture Therapy — Undergo electroacupuncture therapy
  Other Names: Electroacupuncture
  Arms: Group I (electroacupuncture therapy)
Procedure: Electroacupuncture Therapy — Undergo modified electroacupuncture therapy
  Other Names: Electroacupuncture
  Arms: Group II (sham electroacupuncture therapy)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase II trial studies how well electroacupuncture therapy works in reducing chronic pain in patients following surgery for stage I-III breast cancer. Electroacupuncture therapy is a type of complementary integrative medicine in which pulses of weak electrical current are sent through very thin, solid, sterile, stainless steel needles into certain points in the skin. Electroacupuncture therapy may help to lower pain and other surgery-related symptoms.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the initial efficacy of electroacupuncture (EA) in reducing chronic pain in women following treatment for breast cancer.

SECONDARY OBJECTIVES:

I. Determine if EA produces greater improvement in physical functional mobility as compared to sham electroacupuncture (SEA) or waitlist control (WLC)s.

II. Determine if EA produces greater improvement in overall quality of life (QOL) and symptoms related to fatigue, sleep and mood disturbance compared to SEA or WLC.

III. Determine if EA produces lower pain vigilance and awareness as compared to SEA or WLC.

IV. Examine the association between baseline expectancy and outcomes. V. Explore associations between response to acupuncture and biologic measures, including 1) single nucleotide polymorphisms (SNPS) in catechol-O- methyltransferase (COMT) and opioid receptor-mu1 (OPRM1), and 2) autotaxin (ATX)/lysophosphatidic acid (LPA) axis.

VI. Explore if EA reduces emotional, financial, and behavioral concerns among patients and caregivers compared to the SEA or WLC.

OUTLINE: Patients are randomized to 1 of 3 groups.

GROUP I (EA): Patients undergo electroacupuncture therapy over 45 minutes 2-3 times per week over 4 weeks for a total of 10 sessions.

GROUP II (SEA): Patients undergo modified electroacupuncture therapy over 45 minutes 2-3 times per week over 4 weeks for a total of 10 sessions. Acupuncture needles are placed in different locations using a different technique than those used for Group I.

GROUP III (WLC): Patients receive standard of care without any kind of acupuncture therapy.

After completion of study treatment, patients are followed up at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be adult women >/= 18 years of age.
* Be able to read, write, and speak English
* Able to give informed consent
* Have a history of stage I, II, or III breast cancer
* Have a documented visit with an oncologist during the previous 12-months
* Have no current evidence of disease
* Have persistent pain (unrelated to aromatase inhibitors or chemotherapy-induced peripheral neuropathy) for at least 3 months following treatment for breast cancer
* Have pain severity (arithmetic mean of four pain severity items) >= 2 on Brief Pain Inventory (BPI)
* Have worst pain >= to 4 (0-10 numeric rating scale [NRS]) in the preceding week
* Be willing and able to adhere to all study-related procedures
* Have completed all cancer treatment (including surgery, chemotherapy and/or radiation) at least 4 months prior to enrollment
* Have documented lab work with absolute neutrophil count (ANC) >= 1.0 K/uL and platelets >= 50 K/uL in the past 12 months
* If applicable, maintain self-management of lymphedema symptoms being performed at home at time of study entry

Exclusion Criteria:

* Metastatic breast cancer (stage IV)
* Known bleeding disorder per patient reported history
* Cardiac pacemaker or other implanted electronic devices
* New or planned new lymphedema treatment during the study period
* Currently receiving or ever received acupuncture for present pain condition
* Received acupuncture with electrical stimulation for any condition
* Received acupuncture for any condition in the past year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain scores assessed by Brief Pain Inventory (BPI) | Baseline to 8 weeks
  Change in pain scores will be compared between groups. Assessing the initial efficacy of electroacupuncture (EA) relative to sham electroacupuncture (SEA) and waitlist control (WLC), use linear regression and linear mixed model analyses. Pain Scores(0-10) 0 No pain-10 Worst Pain.

SECONDARY OUTCOMES:
Presence of single nucleotide polymorphisms (SNPs) in (COMT) catechol-O- methyltransferase | Up to 8 weeks
  Will explore the correlations between response to acupuncture and presence of different gene variations in (COMT) catechol-O- methyltransferase and (OPRM1). Will use linear regression and linear mixed model analyses.
Presence of single nucleotide polymorphisms (SNPs) in (OPRM1) opioid receptor-mu1 | Up to 8 weeks
  Will explore correlations between response to acupuncture and presence of different gene variations in (COMT) catechol-O- methyltransferase and (OPRM1) opioid receptor-mu1. Will use linear regression and linear mixed model analyses.
Change in autotaxin (ATX)/lysophosphatidic acid (LPA) axis | Baseline to 8 weeks
  Will explore correlations between response to acupuncture and ATX-mediated LPA biosynthesis. Will use linear regression and linear mixed model analyses.
Spouse Behavior Subscale of the Multidimensional Pain Inventory (SBS-MPI) Questionnaire | Up to 8 weeks
  Emotional, financial, and behavioral concerns among patients and caregivers will be compared between (EA) electroacupuncture and (SEA) sham electroacupuncture or (WLC) waitlist control group. (Agree or Disagree 5-1) 1-Strongly Disagree, 2-Disagree, 3-Neither agree or Disagree, 4-Agree 5-Strongly Agree
Caregiver Reaction Assessment (CRA) Questionnaire | Up to 8 weeks
  Emotional, financial, and behavioral concerns among patients and caregivers will be compared between (EA) electroacupuncture and (SEA) sham electroacupuncture or (WLC) waitlist control group. (Agree or Disagree 5-1) 1-Strongly Disagree, 2-Disagree, 3-Neither agree or Disagree, 4-Agree 5-Strongly Agree
Baseline expectancy of participants will be correlated to the outcomes response. | At baseline
  Will use linear regression and linear mixed model analyses.
Physical functional mobility will be compared. | Baseline to 8 weeks
  Change in physical functional mobility will be compared between groups. Assessing the initial efficacy of (EA) electroacupuncture relative to (SEA) sham electroacupuncture and (WLC) waitlist control group., use linear regression and linear mixed model analyses.
Quality of life (QOL) questionnaire | Baseline to 8 weeks
  Change in overall (QOL) Quality of life will be compared between groups. Assessing the initial efficacy of (EA) electroacupuncture relative to (SEA) sham electroacupuncture and (WLC) waitlist control group., use linear regression and linear mixed model analyses.
Changes in symptoms of fatigue questionnaire | Baseline to 8 weeks
  Changes in symptoms of fatigue, sleep, and mood disturbance will be compared between groups. Assessing the initial efficacy of (EA) electroacupuncture (SEA) sham electroacupuncture and (WLC) waitlist control group., use linear regression and linear mixed mode Fatigue (0-10) 0 No Fatigue-10 Fatigue
Changes in symptoms of sleep questionnaire | Baseline to 8 weeks
  Changes in symptoms of fatigue, sleep, and mood disturbance will be compared between groups. Assessing the initial efficacy of (EA) electroacupuncture (SEA) sham electroacupuncture and (WLC) waitlist control group., use linear regression and linear mixed mode. Thee Pittsburgh Sleep Quality Index (PSQI) Very Good (0) Fairly Good (1) Fairly Bad(2) Very Bad (3)
Changes in symptoms of mood disturbance | Baseline to 8 weeks
  Changes in symptoms of fatigue, sleep, and mood disturbance will be compared between groups. Assessing the initial efficacy of (EA) electroacupuncture (SEA) sham electroacupuncture and (WLC) waitlist control group., use linear regression and linear mixed mode. Mood (0-10) 0 Does not interfere, 10 Completely Interferes.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org